CLINICAL TRIAL: NCT00002323
Title: A Multi-Center, Placebo-Controlled, Double-Blind, Randomized Trial Comparing the Virologic and Immunologic Activities of 400 Mg Nevirapine in Combination With Zidovudine Versus Zidovudine Alone in Asymptomatic HIV-1 Infected Patients With 4-12 Months of Prior Zidovudine Therapy and 200-500 CD4+ Cells/mm3
Brief Title: A Multi-Center, Placebo-Controlled, Double-Blind, Randomized Trial Comparing the Virologic and Immunologic Activities of 400 Mg Nevirapine in Combination With Zidovudine Versus Zidovudine Alone in Asymptomatic HIV-1 Infected Patients With 4-12 Months of Prior Zidovudine Therapy and 200-500 CD4+ Cell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 200B; BIPI 1037
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-08

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; Nevirapine
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Zidovudine

INTERVENTIONS:
Drug: Nevirapine
Drug: Zidovudine

SUMMARY:
PRIMARY: To compare the virologic activity (quantitative RNA PCR, quantitative PBMC) of the combination of nevirapine and zidovudine (AZT) versus AZT alone after 3 and 6 months of treatment. To compare the effects of these two regimens on CD4 T-cell count and percentage.

SECONDARY: To compare and evaluate other markers of immunologic and virologic activity in patients receiving nevirapine/AZT versus AZT alone. To compare the effects of the two regimens on clinical signs and symptoms. To evaluate the safety and tolerance of the two regimens.

DETAILED DESCRIPTION:
Patients receive combination nevirapine/AZT or AZT alone. Patients are evaluated for virologic and immunologic activity at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* PCP prophylaxis (trimethoprim-sulfamethoxazole, dapsone, or aerosolized pentamidine), at the discretion of the investigator.
* Antifungal prophylaxis with oral fluconazole or ketoconazole.
* Antiviral prophylaxis for herpes simplex virus with <= 1000 mg/day oral acyclovir.
* Dilantin for prevention and treatment of seizures.

Patients must have:

* Asymptomatic HIV infection.
* CD4 count 200-500 cells/mm3.
* No prior AIDS.
* No history of or active HIV-related thrush, vaginal candidiasis, zoster (shingles), excessive weight loss, persistent fever, or diarrhea.
* Tolerated 500-600 mg AZT daily for at least 4 months but no more than 12 months immediately prior to study entry.
* Consent of parent or guardian if less than 18 years of age.

NOTE:

* Patients may not co-enroll in another protocol involving other investigational drugs or biologics.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Malignancy other than limited cutaneous basal cell carcinoma.
* Psychiatric condition sufficient to impair study compliance.

Concurrent Medication:

Excluded:

* Systemic glucocorticoids and steroid hormones.
* Dicumarol, warfarin, and other anticoagulant medications.
* Cimetidine.
* Tolbutamide.
* Doxycycline.
* Chloramphenicol.
* Phenobarbital and other barbiturates.
* Foscarnet.
* Erythromycin.
* Amoxicillin-clavulanate (Augmentin).
* Ticarcillin clavulanate.
* Biologic response modifiers (alpha interferon, IL-2, immune modulators).
* Any investigational drugs other than study drugs.

Patients with the following prior condition are excluded:

History of clinically important disease other than HIV infection, that may put patient at risk because of participation in this study.

Prior Medication:

Excluded:

* Antiretroviral medications other than AZT.

Excluded within 4 weeks prior to study entry:

* Immunosuppressive or cytotoxic drugs or other experimental drugs.
* Systemic glucocorticoids and steroid hormones.
* Dicumarol, warfarin, and other anticoagulant medications.
* Cimetidine.
* Tolbutamide.
* Doxycycline.
* Chloramphenicol.
* Phenobarbital and other barbiturates.
* Foscarnet.
* Erythromycin.
* Amoxicillin-clavulanate (augmentin).
* Ticarcillin clavulanate.
* Biologic response modifiers (alpha interferon, IL-2, immune modulators).

Required:

* AZT at 500-600 mg/day for at least 4 months but no more than 12 months immediately preceding study entry.

Chronic use of alcohol or drugs sufficient to impair study compliance.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Highland Gen Hosp / San Francisco Gen Hosp, Oakland, California
  - Northwestern Univ Med School, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Washington Univ School of Medicine, St Louis, Missouri
  - Univ TX Galveston Med Branch, Galveston, Texas